Official Title: Using an Internet Survey to Improve Patient Adherence in Chronic Disease

NCT01702883

IRB Approval Date: 07/16/2014



Department of Dermatology

## MEDICATION EXPERIENCE STUDY Informed Consent Form to Participate in Research Steve R Feldman, M.D., Ph.D., Principal Investigator

The survey you are completing is a part of enrollment into a research study of your experience with your medication.

This research study is being done at the Wake Forest Baptist Medical Center (WFBMC) pharmacies recruiting 1112 subjects. The study will evaluate your experience with standard-of-care oral medications used to treat high blood pressure, high cholesterol, diabetes, or depression. The study will last 12 months, via electronic means, by internet or text message access. All subjects are expected to complete several surveys during this time frame.

If you choose to participate, you will automatically move forward to complete the pre-enrollment surveys. It is important to gather baseline information; therefore all subjects need to complete the pre-enrollment survey. In order to understand experiences over time, subjects will be complete additional surveys during the 12 months. We will send you an email or text message invitation to log-on to the survey website or by other electronic means (such as smart phone or text message) when it is time to complete another survey. You will click a link in the email or text message that will take you directly to the survey website, where you will share your experiences with your medicines. The survey will ask just a few short, simple questions about your experience with your medication. It will contain questions on how many times the medication was used, how easy or difficult it was to take, how helpful it was, and what side effects were experienced.

Please notify the investigator and discontinue study enrollment if you are told by your physician to stop taking the medication being studied before the end of the study, or if you must stop using the WFBMC pharmacy to obtain the medication. The investigator also has the right to stop your participation in the study at any time. This could be because new information becomes available, you failed to follow instructions, or because the entire study has been stopped.

You will be given any new information we become aware of that would affect your willingness to continue to participate in the study.

Taking part in this research study may involve providing information that you consider confidential or private. Efforts will be made to keep the information about your medications confidential and not shared with anyone not involved in this study. The answers to the surveys will also be kept confidential, in password protected electronic files. If you experience any side effects after taking your medicine, then you should discuss them with the doctor that prescribed your medicine.

Taking part in this study is voluntary. You may choose not to take part or you may leave the study at any time. Refusing to participate or leaving the study will not affect your current or future care at WFUHS. You may drop out at any time, please let the study staff know that you no longer intend to participate. By completing the survey, you are implying consent to participate in this research study.

You will receive an entry each month you are actively in the study for a quarterly drawing to win an iPad mini.

Wake Forest University Health Sciences has applied for a patent for the electronic survey program and may start a company to sell it. In this case, the medical school and Dr. Feldman will hold stock in the company and may receive income from its sales. The medical school and Dr. Feldman also hold stock in the company that will provide the data management.

| For questions about the study of | contact the study investigator, Steven R. Feldman, M.D., Ph.D. at | or via email |
|---|---|---|
| at | or The Institutional Review Board (IRB) is a group of people who review th | ne research to |
| protect your rights. If you ha | ave a question about your rights as a research participant, or you would lil | ke to discuss |
| problems or concerns, have q | juestions or want to offer input, or you want to obtain additional information | ı, you should |
| contact the Chairman of the IR | RB at | |

You can print a copy of this document for your records or have it emailed to you to print at a later time.

Page 1 of 1

Version: